CLINICAL TRIAL: NCT06406582
Title: Surface Conditioning Effectiveness, Accuracy and Treatment Result of Zirconia Laminate Veneer
Brief Title: Treatment Result of Zirconia Laminate Veneer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01050122106
Record Dates: First submitted 2024-05-03; First posted 2024-05-09 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-05

CONDITIONS: Dislocation, Tooth; Teeth, Endodontically-Treated; Tooth Fracture; Tooth Injuries; Tooth Abnormalities; Cracked Tooth Syndrome; Tooth Crowding
Keywords: ceramic laminate veneers; zirconia; lithium disilicate; computer-aided manufacturing
MeSH Terms: conditions — Tooth Avulsion; Tooth, Nonvital; Tooth Fractures; Tooth Injuries; Tooth Abnormalities; Cracked Tooth Syndrome; Malocclusion

STUDY DESIGN:
Intervention Model Description: Zirconia Group (Intervention): Participants receive zirconia laminate veneers. Lithium Disilicate Group (Control): Participants receive lithium disilicate laminate veneers. Lithium disilicate is a standard ceramic material for laminate veneers.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind. Both participants and the outcomes assessor are kept unaware of which ceramic laminate veneer material (Zirconia or Lithium Disilicate) the participants are receiving
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zirconia laminate veneer (Experimental): Intervention: Single-tooth restoration using zirconia ceramic laminate veneers.
  Procedure:
  Tooth preparation following standard protocols for laminate veneer placement. Fabrication of zirconia laminate veneers. Cementation of zirconia laminate veneers with appropriate bonding protocol. Follow-Up: after 2 weeks, 6 months, and 12 months
  Interventions: Device: Zirconia laminate veneer
- Lithium Disilicate laminate veneer (Active Comparator): Intervention: Single-tooth restoration using lithium disilicate ceramic laminate veneers.
  Procedure:
  Tooth preparation following standard protocols for laminate veneer placement. Fabrication of lithium disilicate laminate veneers. Cementation of lithium disilicate laminate veneers with appropriate bonding protocol.
  Follow-Up: after 2 weeks, 6 months, and 12 months
  Interventions: Device: Lithium Disilicate laminate veneer

INTERVENTIONS:
Device: Zirconia laminate veneer — Zirconia veneers are milled with computer-aided manufacturing technology from multilayered zirconia discs with shade matched with adjacent teeth. After sintering, veneer surfaces are treated with a hydrofluoric acid-nitric acid mixture. Next, veneers are cut back if necessary to provide space for characterization. Veneers are bonded with a light-cured veneer adhesive system (Relyx Veneer LC, 3M, USA).
  Arms: Zirconia laminate veneer
Device: Lithium Disilicate laminate veneer — Lithium Disilicate veneers are milled with computer-aided manufacturing technology from lithium disilicate blocks with shade matched with adjacent teeth. After sintering, veneer surfaces are treated with hydrofluoric acid. Next, veneers are cut back if necessary to provide space for characterization. Veneers are bonded with a light-cured veneer adhesive system (Relyx Veneer LC, 3M, USA).
  Arms: Lithium Disilicate laminate veneer

SUMMARY:
This study aims to evaluate the clinical performance of the zirconia laminate veneer, a minimally invasive prosthetic restoration

DETAILED DESCRIPTION:
Patients with indications for single tooth restoration with ceramic laminate veneers are recruited for the study. These indications include spaced, discolored, malformed, root canal-treated, chipped, and mildly crowded teeth. After providing written informed consent, all patients are randomly divided into two groups in a double-blind manner (participants and the outcomes assessor) in a 1:1 ratio, including the Zirconia group (intervention) and the Lithium Disilicate group (control). Each patient's tooth is prepared and restored with the corresponding laminate veneer material, that is, zirconia and lithium disilicate.

ELIGIBILITY:
Inclusion Criteria:

* Spaced tooth
* Discolored tooth
* Malformed tooth
* Root canal-treated tooth
* Chipped tooth
* Mildly crowded tooth

Exclusion Criteria:

* Tooth bruxism
* Inadequate enamel for bonding
* Large restoration exists
* Bad oral habits harming restoration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Marginal and internal fit | Before veneer adhesion
  Measurement of marginal and internal fit in micrometers with silicone replica method
Gingival health | 2 weeks, 6 months, 12 months
  Assessment of gingival index
Periodontal pocket | 2 weeks, 6 months, 12 months
  Measurement of periodontal pocket depth in millimeters
Evaluation criteria based on the modified United States Public Health Standard | 2 weeks, 6 months, 12 months
  Shade match, contour, fracture, loss of retention, hypersensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- High Technical Center of Dentistry, School of Dentistry, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No